CLINICAL TRIAL: NCT02956057
Title: A Head-to-head Comparison of Efficiency and Tolerance of 4-L Polyethylene Glycol and Sodium Picosulphate/ Magnesium Citrate, Polyethylene Glycol/Ascorbate Before Colonoscopy
Brief Title: Polyethylene Glycol Versus Low Volume Solutions Prior to Colonoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tomas Bata Hospital, Czech Republic (Other)
Collaborators: Brno University Hospital (Other); Faculty Hospital Kralovske Vinohrady (Other Government)
Responsible Party: Principal Investigator, Vladimir Kojecky, MD, Ph.D., MUDr., Tomas Bata Hospital, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BN102016
Record Dates: First submitted 2016-11-01; First posted 2016-11-04 (Estimated); Results first posted 2020-10-28 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Colonoscopy
MeSH Terms: interventions — Polyethylene Glycols; magnesium citrate; Ascorbic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- PEG1D (Active Comparator): Polyethylene glycols single dose a day before colonoscopy
  Interventions: Drug: Polyethylene Glycols
- PEG2D (Active Comparator): Polyethylene glycols split dose
  Interventions: Drug: Polyethylene Glycols
- SPMC1D (Active Comparator): Natrium picosulfate/ Magnesium citrate single dose day before colonoscopy
  Interventions: Drug: Natrium picosulfate / Magnesium citrate
- SPMC2D (Active Comparator): Natrium picosulfate/ Magnesium citrate split dose
  Interventions: Drug: Natrium picosulfate / Magnesium citrate
- PEGA1D (Active Comparator): Polyethylene glycol / Ascorbic acid single dose day before colonoscopy
  Interventions: Drug: Polyethylene glycol / Ascorbic acid
- PEGA2D (Active Comparator): Polyethylene glycol / Ascorbic acid split dose
  Interventions: Drug: Polyethylene glycol / Ascorbic acid

INTERVENTIONS:
Drug: Polyethylene Glycols
  Arms: PEG1D; PEG2D
Drug: Natrium picosulfate / Magnesium citrate
  Arms: SPMC1D; SPMC2D
Drug: Polyethylene glycol / Ascorbic acid
  Arms: PEGA1D; PEGA2D

SUMMARY:
Study evaluates the efficacy and tolerability of low volume preparations compared with conventional 4L polyethylene glycol prior to colonoscopy

DETAILED DESCRIPTION:
To compare the efficacy and tolerance of standard polyethylene glycol to low volume sodium picosulphate/magnesium citrate and polyethylene glycol/ascorbic acid in a single or split dose regimen for colonoscopy bowel preparation in a head-to-head design.

ELIGIBILITY:
Inclusion Criteria:

* Subjects referred to diagnostic or therapeutic colonoscopy

Exclusion Criteria:

* ileus
* known or suspected bowel obstruction
* active bowel inflammation
* pregnancy
* any presence of serious medical conditions
* history of prior colonic or rectal surgery
* inability to obtain valid data from subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1044 (Actual)
Dates: Start 2016-11-12 (Actual); Primary Completion 2017-05-29 (Actual); Study Completion 2017-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Kojecky, MD, Principal Investigator — Nemocnice T.Bati
Locations (1):
- Faculty Hospital Kralovske Vinohrady, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kojecky V, Matous J, Keil R, Dastych M, Kroupa R, Zadorova Z, Varga M, Dolina J, Kment M, Hep A. A head-to-head comparison of 4-L polyethylene glycol and low-volume solutions before colonoscopy: which is the best? A multicentre, randomized trial. Int J Colorectal Dis. 2017 Dec;32(12):1763-1766. doi: 10.1007/s00384-017-2901-x. Epub 2017 Sep 24. PMID 28944412

RESULTS

PARTICIPANT FLOW:
Groups:
- PEG1D: Polyethylene glycols single dose a day before colonoscopy
  Polyethylene Glycols
- PEG2D: Polyethylene glycols split dose
  Polyethylene Glycols
- SPMC1D: Natrium picosulfate/ Magnesium citrate single dose day before colonoscopy
  Natrium picosulfate / Magnesium citrate
- SPMC2D: Natrium picosulfate/ Magnesium citrate split dose
  Natrium picosulfate / Magnesium citrate
- PEGA1D: Polyethylene glycol / Ascorbic acid single dose day before colonoscopy
  Polyethylene glycol / Ascorbic acid
- PEGA2D: Polyethylene glycol / Ascorbic acid split dose
  Polyethylene glycol / Ascorbic acid
Period: Overall Study
Arm/Group | PEG1D | PEG2D | SPMC1D | SPMC2D | PEGA1D | PEGA2D
Started | 174 | 174 | 174 | 174 | 174 | 174
Completed | 160 | 162 | 166 | 159 | 169 | 157
Not Completed | 14 | 12 | 8 | 15 | 5 | 17
Not completed — Discontinued intervention | 14 | 10 | 7 | 14 | 4 | 17
Not completed — Lost to Follow-up | 0 | 2 | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PEG1D | PEG2D | SPMC1D | SPMC2D | PEGA1D | PEGA2D | Total
Number analyzed (Participants) | 160 | 162 | 166 | 159 | 169 | 157 | 973
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (15.3) | 64.5 (13.9) | 60.8 (16.1) | 63.1 (13.1) | 60.1 (14.3) | 60.6 (17.0) | 62.1 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 70 | 81 | 77 | 67 | 67 | 429
  Male | 93 | 92 | 85 | 82 | 102 | 90 | 544
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 160 | 162 | 166 | 159 | 169 | 157 | 973
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Czechia | 160 | 162 | 166 | 159 | 169 | 157 | 973

OUTCOME MEASURES:

1. Primary Outcome: Quality of Bowel Preparation Using the Aronchick Scale ( Score 1+2)
Description: Bowel preparation score 1+2 expressed on Aronchick scale (1 the best, 5 the worst)
Time Frame: One day
Measure: Count of Participants; unit: Participants
Arm/Group | PEG1D | PEG2D | SPMC1D | SPMC2D | PEGA1D | PEGA2D
Number analyzed (Participants) | 160 | 162 | 166 | 159 | 169 | 157
Participants | 110 | 145 | 100 | 134 | 121 | 55

2. Secondary Outcome: Tolerance of Bowel Preparation Assessed by 5 Point VAS ( Score 1+2)
Description: Tolerance of Bowel Preparation Assessed by VAS score 1+2 ( 1-excellent, 5-very poor)
Time Frame: One day
Measure: Count of Participants; unit: Participants
Arm/Group | PEG1D | PEG2D | SPMC1D | SPMC2D | PEGA1D | PEGA2D
Number analyzed (Participants) | 160 | 162 | 166 | 159 | 169 | 157
Participants | 56 | 72 | 134 | 139 | 85 | 80

ADVERSE EVENTS:
Time Frame: 0
Description: AE not assessed
Arm/Group | PEG1D | PEG2D | SPMC1D | SPMC2D | PEGA1D | PEGA2D
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-03): https://cdn.clinicaltrials.gov/large-docs/57/NCT02956057/Prot_SAP_000.pdf